CLINICAL TRIAL: NCT03696901
Title: Xydalba Utilization Registry: A Multicenter, Prospective and Retrospective Registry to Characterize the Use of Xydalba
Brief Title: Xydalba Utilization Registry in Germany
Status: Terminated | Type: Observational
Why Stopped: Terminated
Sponsor: Correvio International Sarl (Industry)
Collaborators: AMS Advanced Medical Services GmbH (Industry); PrimeVigilance (Industry)
Responsible Party: Sponsor
Organization: Advanz Pharma (Industry)
Other Study IDs: DAL-REG01-GER
Record Dates: First submitted 2018-05-09; First posted 2018-10-05 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Bacterial Infections
Keywords: Dalbavancine; Xydalba
MeSH Terms: conditions — Bacterial Infections | interventions — dalbavancin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- use of Xydalba, >18 years: Male and female patients, ≥18 years of age at the time of receipt of Xydalba. Patients who received at least one Xydalba administration in Germany
  Interventions: Drug: Xydalba

INTERVENTIONS:
Drug: Xydalba — Information will be recorded about Xydalba administration (e.g. dose(s), number of infusions, length of infusions, dates or schedule of administration, sites of administration [e.g. hospital, ICU]), and reason for discontinuation, including response to treatment to assess whether the patient was clinically improving when Xydalba was discontinued
  Other Names: Dalbavancin

SUMMARY:
This observational study will collect data on the use of the drug Xydalba® in daily clinical practice in Germany. Such observational studies are also referred to as registries. The sponsor of the study is Correvio International Sárl, based in Switzerland.

Xydalba® contains the active substance dalbavancin, a remedy for a certain type of bacterial pathogens (so-called "gram positive bacteria") which cause the disease. Active ingredients against bacteria are also called antibiotics.

Correvio wants to know which patients received the drug and how the disease went. The treatment places where you got Xydalba, ie clinic, intensive care unit or elsewhere should be recorded. In addition, it is important in this type of medication to track whether the pathogens are changing in any way. Any safety-relevant events (such as side effects) that have occurred during treatment should be investigated by the sponsor and submitted to the competent European authorities.

DETAILED DESCRIPTION:
OBJECTIVES

The objectives of this registry are as follows:

* To determine the following characteristics in patients who received intravenous Xydalba administration:

  * Patient characteristics.
  * Disease characteristics.
  * Pathogen characteristics.
* To characterize the usage of Xydalba.
* To characterize the patient's residence and, in hospitalized patients, the lengths of hospital and intensive care unit (ICU) stays, and the destination upon hospital discharge.
* To assess the response of Xydalba treatment, based on clinician determination.
* To characterize the major healthcare resource utilization (HRU) of patients treated with Xydalba.

REGISTRY DESIGN This is a multicenter, prospective and retrospective registry of adult patients treated with Xydalba in Germany.

All Adverse events (AEs) (serious and non-serious; special situations; related and not-related, collected prospectively or retrospectively) will be recorded in the eCRF. Treatment related AEs and SAEs will be reported to the healthcare authorities, as requested by local regulations and according to current Guideline on good pharmacovigilance practices (GVP) Module VI - Collection, management and submission of reports of suspected adverse reactions to medicinal products (Rev 2).

TEST PRODUCT (S), DOSE, AND MODE OF ADMINISTRATION Xydalba (dalbavancin) as prescribed by the physician according to clinical practice.

RATIONALE This prospective and retrospective registry is designed to capture information about the clinical use of Xydalba, its safety and effectiveness, characteristics of the patient, disease, pathogen, clinical course, treatment course, and hospitalization. This registry will capture the data in real world setting on patients who received Xydalba.

ELIGIBILITY:
Inclusion Criteria A patient must meet all of the following criteria to be eligible for participation in the study.

1. Male and female patient, ≥18 years of age at the time of receipt of Xydalba.
2. The patient received at least one infusion of Xydalba.
3. Patient signed the consent form

Exclusion Criteria A patient who meets the following criterion is not eligible for participation in the study.

1. The patient was enrolled in a clinical trial in which treatment for Xydalba is managed through a protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will capture the data in real world setting on patients who received at least one does of Xydalba.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of ABSSSI and other primary diagnoses among patients who received Xydalba (dalbavancin) as treatment for this primary diagnosis | Day of first dose

SECONDARY OUTCOMES:
Clinical response | at 30 days after first dose
  Clinical response by cured, improved, failure, non-evaluable, worsening or other (non-clinically evaluable)
Clinical response by diagnosis | at 30 days after first dose
  Clinical response by diagnosis (ABSSSI, Gram-positive bacteremia, other associated diagnosis)
Time from Xydalba treatment onset to clinical response | up to 30 days after first dose
Adverse Events, Adverse Drug Reactions and Special Situations | up to 30 days after first dose

OTHER OUTCOMES:
Xydalba Treatment dose(s) | up to 30 days after first dose
  Dose(s) of Xydalba in mg per infusion
Number of Xydalba Infusions | up to 30 days after first dose
  number of Infusions given
Length of Xydalba Infusions | up to 30 days after first dose
  length of Infusions in minutes
Days of Xydalba treatment | up to 30 days after first dose
  number of Days of treatment
Percentage of monotherapy vs. concurrent therapy | up to 30 days after first dose
  % of cases for which Xydalba is given as monotherapy and % of cases for which Xydalba is given as concurrent therapy
Percentage first-line vs. subsequent-line monotherapy | up to 30 days after first dose
  % of cases for which Xydalba is given as first-line and % of cases for which Xydalba is given as subsequent-line
Prior Antibiotic Therapies | from the time of the primary specified infectious disease diagnosis until Xydalba treatment (estimated to be within 3 months of Xydalba treatment)
  Descriptive summary of other antibiotic therapies received
Reason for discontinuation | up to 30 days after first dose
  descriptive listing of type of reasons

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Bhirangi, MBBS FRCS I, Study Director — Correvio International Sarl
Locations (7):
- Germany (7):
  - Universitätsklinikum Essen / Klinik für Infektiologie, Essen
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Universitätsklinikum Jena, Jena
  - Klinikum der Universität München / Klinische Mikrobiologie und Krankenhaushygiene, München
  - Universitätsklinikum Regensburg /Stabsstelle Infektiologie, Regensburg
  - Universitätsklinikum Rostock Abteilung für Tropenmedizin und Infektionskrankheiten Zentrum für Innere Medizin, Rostock

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ventola CL. The antibiotic resistance crisis: part 1: causes and threats. P T. 2015 Apr;40(4):277-83. PMID 25859123
- [Background] Garau J, Ostermann H, Medina J, Avila M, McBride K, Blasi F; REACH study group. Current management of patients hospitalized with complicated skin and soft tissue infections across Europe (2010-2011): assessment of clinical practice patterns and real-life effectiveness of antibiotics from the REACH study. Clin Microbiol Infect. 2013 Sep;19(9):E377-85. doi: 10.1111/1469-0691.12235. Epub 2013 May 10. PMID 23663184
- [Background] Morbidité et mortalité des infections à bactéries multi-résistantes aux antibiotiques en France en 2012. Étude Burden BMR, rapport - Juin 2015. Saint-Maurice : Institut de veille sanitaire ; 2015. 21p. Disponible à partir de l'URL : http://www.invs.sante.fr
- [Background] Rolain JM, Abat C, Jimeno MT, Fournier PE, Raoult D. Do we need new antibiotics? Clin Microbiol Infect. 2016 May;22(5):408-15. doi: 10.1016/j.cmi.2016.03.012. Epub 2016 Mar 26. PMID 27021418
- [Background] EMA Assessment Report 2015. http://www.ema.europa.eu/docs/en_GB/document_library/EPAR_-_Public_assessment_report/human/002840/WC500183871.pdf
- [Background] Smith JR, Roberts KD, Rybak MJ. Dalbavancin: A Novel Lipoglycopeptide Antibiotic with Extended Activity Against Gram-Positive Infections. Infect Dis Ther. 2015 Sep;4(3):245-58. doi: 10.1007/s40121-015-0077-7. Epub 2015 Sep 4. PMID 26341488
- [Background] Xydalba approval history. Drugs.com. http://www.drugs.com/history/Xydalba.html. Accessed February 3, 2016
- [Background] Boucher HW, Wilcox M, Talbot GH, Puttagunta S, Das AF, Dunne MW. Once-weekly dalbavancin versus daily conventional therapy for skin infection. N Engl J Med. 2014 Jun 5;370(23):2169-79. doi: 10.1056/NEJMoa1310480. PMID 24897082
- [Background] Guideline on good pharmacovigilance practices (GVP) Module VI - Collection, management and submission of reports of suspected adverse reactions to medicinal products
- Available data/document: Study Protocol: Xydalba — https://awbdb.bfarm.de/ords/f?p=101:STARTSEITE:::::: — BfArM AWB Datenbank